CLINICAL TRIAL: NCT07076121
Title: A Randomized, Phase 2/3 Study Comparing BMS-986504 in Combination With Nab-paclitaxel and Gemcitabine Versus Placebo in Combination With Nab-paclitaxel and Gemcitabine in Participants With Untreated Metastatic Pancreatic Ductal Adenocarcinoma Harboring Homozygous MTAP Deletion
Brief Title: A Study Comparing BMS-986504 in Combination With Nab-paclitaxel and Gemcitabine Versus Placebo in Combination With Nab-paclitaxel and Gemcitabine in Participants With Untreated Metastatic Pancreatic Ductal Adenocarcinoma With Homozygous MTAP Deletion (MountainTAP-30)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA240-0030; 2025-522598-12 (Other: EU CTR); U1111-1320-4708 (Other: WHO); CA2400030 (Other: Bristol-Myers Squibb Protocol ID)
Record Dates: First submitted 2025-07-14; First posted 2025-07-21 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: PRMT5; MTAP; MRTX1719; MountainTAP; Pancreatic cancer; PDAC
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Arm A (Experimental)
  Interventions: Drug: BMS-986504; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Arm B (Experimental)
  Interventions: Drug: BMS-986504; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Arm C (Placebo Comparator)
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Placebo
- Arm D (Placebo Comparator)
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Placebo
- Arm E (Experimental)
  Interventions: Drug: BMS-986504; Drug: Gemcitabine; Drug: Nab-paclitaxel
- Arm F (Placebo Comparator)
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: BMS-986504 — Specified dose on specified days
  Other Names: MRTX1719
  Arms: Arm A; Arm B; Arm E
Drug: Gemcitabine — Specified dose on specified days
Drug: Nab-paclitaxel — Specified dose on specified days
  Other Names: Abraxane
Drug: Placebo — Specified dose on specified days
  Arms: Arm C; Arm D; Arm F

SUMMARY:
The purpose of this study is to assess the safety and efficacy of BMS-986504, a selective, MTA-cooperative PRMT5 inhibitor, in combination with Nab-paclitaxel/Gemcitabine (nab-p/gem) versus placebo in combination with nab-p/gem, in participants with untreated metastatic Pancreatic Ductal Adenocarcinoma (PDAC) with homozygous methylthioadenosine phosphorylase (MTAP) deletion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic pancreatic ductal adenocarcinoma (PDAC).
* Evidence of homozygous methylthioadenosine phosphorylase (MTAP) deletion or MTAP loss detected in tumor tissue.
* Metastatic disease with at least 1 measurable lesion as per Response Evaluation Criteria in Solid Tumors version v1.1 (RECIST v1.1).
* Participants must not have received any systemic anticancer treatments in the metastatic setting.
* If clinically indicated and as per investigator discretion, participants may receive up to 1 cycle of Nab-paclitaxel/Gemcitabine (nab-p/gem) in the metastatic setting and must have not progressed or required discontinuation due to intolerable toxicity.
* Initial cycle of nab-p/gem administered in the metastatic setting must have been completed prior to randomization.

Exclusion Criteria:

* Concurrent malignancy (present during screening) requiring treatment or history of prior malignancy active within 2 years prior to screening.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 470 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2029-05-03 (Estimated); Study Completion 2029-05-03 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival as assessed by Response Evaluation Criteria in Solid Tumors version v1.1 (RECIST v1.1) | Up to 3 years after last participant is randomized
  Defined as the time between the randomization date and the date of progressive disease (PD) or death from any cause (whichever occurs first)
Overall Survival (OS) | Up to 3 years after last participant is randomized
  Defined as the time from the randomization date to the date of death from any cause

SECONDARY OUTCOMES:
Objective Response (OR) as assessed by RECIST v1.1 | Up to 3 years after last participant is randomized
Duration of Response (DOR) as assessed by RECIST v1.1 | Up to 3 years after last participant is randomized
  Defined as the time between the date of the first documentation of objective tumor response (complete response (CR) or partial response (PR)) and the date of disease progression or to death from any cause (whichever occurs first)
Time to Objective Response (TTOR) as assessed by RECIST v1.1 | Up to 3 years after last participant is randomized
  Defined as the time between randomization to the date of the first documentation of objective tumor response
Disease control as assessed by RECIST v1.1 | Up to 3 years after last participant is randomized
  Defined as the best overall response (BOR) of confirmed CR, PR, or stable disease (SD)
PFS as assessed by RECIST v1.1 | Up to 3 years after last participant is randomized

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (275):
- United States (48):
  - Local Institution - 0142, Phoenix, Arizona
  - Local Institution - 0365, Tucson, Arizona
  - Highlands Oncology Group, Springdale, Arkansas
  - Local Institution - 0373, La Jolla, California
  - Local Institution - 0157, San Francisco, California
  - Local Institution - 0369, Jacksonville, Florida
  - Local Institution - 0139, Jacksonville, Florida
  - Local Institution - 0132, Tampa, Florida
  - Local Institution - 0367, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - St. Luke's Cancer Institute: Boise, Boise, Idaho
  - Local Institution - 0168, Chicago, Illinois
  - Local Institution - 0125, Westwood, Kansas
  - Local Institution - 0370, Louisville, Kentucky
  - Local Institution - 0371, Baltimore, Maryland
  - Local Institution - 0145, Baltimore, Maryland
  - Local Institution - 0120, Boston, Massachusetts
  - Local Institution - 0191, Detroit, Michigan
  - The Cancer & Hematology Centers, Grand Rapids, Michigan
  - Local Institution - 0182, Rochester, Minnesota
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - Local Institution - 0144, Buffalo, New York
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Local Institution - 0377, Mineola, New York
  - Local Institution - 0143, New York, New York
  - Local Institution - 0140, New York, New York
  - Local Institution - 0279, New York, New York
  - Local Institution - 0161, Rochester, New York
  - Local Institution - 0129, Chapel Hill, North Carolina
  - Local Institution - 0376, Columbus, Ohio
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Local Institution - 0162, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Local Institution - 0301, Lancaster, Pennsylvania
  - Local Institution - 0158, Philadelphia, Pennsylvania
  - Local Institution - 0368, Pittsburgh, Pennsylvania
  - Local Institution - 0289, Pittsburgh, Pennsylvania
  - Local Institution - 0167, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - DFW, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Local Institution - 0170, Temple, Texas
  - Local Institution - 0344, Salt Lake City, Utah
  - Local Institution - 0159, Fairfax, Virginia
  - Local Institution - 0348, Norfolk, Virginia
  - Local Institution - 0169, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Local Institution - 0195, Milwaukee, Wisconsin
- Argentina (6):
  - Hospital Británico de Buenos Aires, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 0044, ABB, Buenos Aires F.D.
  - Clínica Mayo de Urgencias Médicas Cruz Blanca S.R.L, San Miguel de Tucumán, Tucumán Province
  - Centro de Educación Médica e Investigaciones clínicas "Dr. Norberto Quirno" (CEMIC), Buenos Aires
  - Sanatorio Allende - Nueva Córdoba, Córdoba
- Australia (7):
  - GenesisCare North Shore, St Leonards, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Local Institution - 0226, Brisbane, Queensland
  - Local Institution - 0229, Woodville, South Australia
  - Cabrini Hospital - Malvern, Malvern, Victoria
  - Local Institution - 0231, Melbourne, Victoria
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (3):
  - Ordensklinikum Linz, Linz, Upper Austria
  - Uniklinikum Salzburg, Salzburg
  - Local Institution - 0211, Vienna
- Belgium (7):
  - Local Institution - 0031, Bonheiden, Antwerpen
  - Local Institution - 0035, Edegem, Antwerpen
  - Local Institution - 0065, Brussels, Bruxelles-Capitale, Région de
  - Local Institution - 0063, Brussels, Bruxelles-Capitale, Région de
  - Local Institution - 0033, Ghent, Oost-Vlaanderen
  - Local Institution - 0032, Leuven, Vlaams-Brabant
  - Local Institution - 0034, Liège
- Brazil (9):
  - Local Institution - 0102, Vitória, Espírito Santo
  - Local Institution - 0291, Salvador, Estado de Bahia
  - Local Institution - 0101, Belo Horizonte, Minas Gerais
  - Local Institution - 0074, Natal, Rio Grande do Norte
  - Local Institution - 0104, Santa Cruz do Sul, Rio Grande do Sul
  - Local Institution - 0071, Barretos, São Paulo
  - Local Institution - 0100, Rio de Janeiro
  - Local Institution - 0075, São Paulo
  - Local Institution - 0332, São Paulo
- Canada (6):
  - Local Institution - 0199, Calgary, Alberta
  - Local Institution - 0200, Vancouver, British Columbia
  - Local Institution - 0202, Halifax, Nova Scotia
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Chile (4):
  - Local Institution - 0156, Viña del Mar, Región de Valparaíso
  - Local Institution - 0048, Santiago, Santiago Metropolitan
  - Local Institution - 0046, Santiago, Santiago Metropolitan
  - Local Institution - 0047, Santiago, Santiago Metropolitan
- China (32):
  - Local Institution - 0312, Hefei, Anhui
  - Local Institution - 0331, Hefei, Anhui
  - Local Institution - 0346, Beijing, Beijing Municipality
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Local Institution - 0307, Chongqing, Chongqing Municipality
  - Local Institution - 0296, Fuzhou, Fujian
  - Local Institution - 0297, Fuzhou, Fujian
  - Local Institution - 0352, Guangzhou, Guangdong
  - Local Institution - 0313, Guangzhou, Guangdong
  - Local Institution - 0302, Harbin, Heilongjiang
  - Local Institution - 0295, Luoyang, Henan
  - Local Institution - 0353, Zhengzhou, Henan
  - Local Institution - 0357, Wuhan, Hubei
  - Local Institution - 0298, Wuhan, Hubei
  - Local Institution - 0293, Changsha, Hunan
  - Local Institution - 0354, Changzhou, Jiangsu
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - Local Institution - 0311, Nanjing, Jiangsu
  - Local Institution - 0304, Shenyang, Liaoning
  - Local Institution - 0345, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Local Institution - 0334, Jining, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Local Institution - 0355, Shanghai, Shanghai Municipality
  - Local Institution - 0300, Shanghai, Shanghai Municipality
  - Local Institution - 0239, Shanghai Shi, Shanghai Municipality
  - Local Institution - 0351, Taiyuan, Shanxi
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - Local Institution - 0305, Chengdu, Sichuan
  - Tianjin Tumor Hospital, Tianjin, Tianjin Municipality
  - Local Institution - 0356, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Colombia (6):
  - Local Institution - 0267, Medellín, Antioquia
  - Local Institution - 0338, Rionegro, Antioquia
  - Local Institution - 0362, Rionegro, Antioquia
  - Local Institution - 0269, Montería, Departamento de Córdoba
  - Local Institution - 0268, Pereira, Risaralda Department
  - Local Institution - 0266, Bogotá
- Czechia (6):
  - Local Institution - 0057, Brno, Brno-město
  - Local Institution - 0060, Hradec Králové, Hradec Králové
  - Local Institution - 0070, Olomouc, Olomoucký kraj
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Local Institution - 0119, Prague, Praha 5
  - Local Institution - 0130, Prague
- Denmark (5):
  - Local Institution - 0019, Copenhagen, Capital Region
  - Local Institution - 0116, Aarhus, Central Jutland
  - Local Institution - 0021, Aalborg, North Denmark
  - Local Institution - 0020, Odense, Region Syddanmark
  - Vejle Sygehus, Vejle, Region Syddanmark
- France (14):
  - Local Institution - 0067, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand, Auvergne
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - Local Institution - 0062, Besançon, Doubs
  - CHU Rangueil, Toulouse, Haute-Garonne
  - Local Institution - 0068, Saint-Cloud, Hauts-de-Seine
  - Local Institution - 0029, Montpellier, Hérault
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de la Côte Basque, Bayonne, Pyrénées-Atlantiques
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Local Institution - 0066, Poitiers, Vienne
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Universitaire Paul Brousse, Villejuif
- Germany (10):
  - Local Institution - 0242, München, Bavaria
  - Krankenhaus Nordwest GmbH, Frankfurt am Main, Hesse
  - Universitätsmedizin Göttingen - Georg-August-Universität, Göttingen, Lower Saxony
  - Local Institution - 0205, Bochum, North Rhine-Westphalia
  - Klinikum Chemnitz - Flemmingstraße, Chemnitz, Saxony
  - Local Institution - 0224, Dresden, Saxony
  - DRK Kliniken Berlin - Köpenick, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Facharztzentrum Eppendorf, Hamburg
  - Universitaetsklinikum Ulm, Ulm
- Greece (7):
  - Local Institution - 0085, Athens, Attikí (Region)
  - Local Institution - 0086, Athens, Attikí (Region)
  - Local Institution - 0084, Athens, Attikí
  - Local Institution - 0259, Heraklion, Irakleío
  - Local Institution - 0091, Thessaloniki, Kentrikí Makedonía
  - Local Institution - 0082, Thessaloniki, Thessaloníki
  - Local Institution - 0083, Larissa, Thessalía
- Hong Kong (2):
  - Local Institution - 0271, Hong Kong
  - Local Institution - 0270, Shatin
- India (7):
  - Local Institution - 0188, Kochi, Kerala
  - Local Institution - 0152, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0179, Bhubaneswar, Odisha
  - Local Institution - 0190, Hyderabad, Telangana
  - Local Institution - 0147, Hyderabad, Telangana
  - Local Institution - 0154, Varanasi, Uttar Pradesh
  - Local Institution - 0153, Kolkata, West Bengal
- Local Institution - 0225, Dublin, Ireland
- Israel (6):
  - Local Institution - 0078, Ramat Gan, Central District
  - Local Institution - 0080, Ẕerifin, Central District
  - Local Institution - 0097, Jerusalem, Jerusalem
  - Local Institution - 0077, Afula, Northern District
  - Local Institution - 0076, Tel Aviv, Tell Abīb
  - Local Institution - 0081, Petah Tikva
- Italy (9):
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - Local Institution - 0092, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Local Institution - 0093, Padua, Veneto
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona
- Japan (7):
  - Local Institution - 0222, Nagoya, Aichi-ken
  - Local Institution - 0217, Kashiwa, Chiba
  - Local Institution - 0219, Sapporo, Hokkaido
  - Local Institution - 0218, Yokohama, Kanagawa
  - Local Institution - 0216, Chuo-ku, Tokyo
  - Local Institution - 0220, Koto, Tokyo
  - Local Institution - 0221, Osaka
- Malaysia (3):
  - Local Institution - 0258, Kuala Lumpur, Kuala Lumpur
  - Local Institution - 0256, Lembah Pantai, Kuala Lumpur
  - Local Institution - 0257, Kuching, Sarawak
- Mexico (9):
  - Local Institution - 0364, Zapopan, Jalisco
  - Local Institution - 0261, Cuauhtémoc, Ciudad de México, Mexico City
  - Local Institution - 0260, Mexico City, Mexico City
  - Local Institution - 0264, Monterrey, Nuevo León
  - Local Institution - 0265, Oaxaca City, Oaxaca
  - Local Institution - 0281, Querétaro City, Querétaro
  - Local Institution - 0372, Mérida, Yucatán
  - Local Institution - 0263, Mexico City
  - Local Institution - 0262, Puebla City
- Netherlands (4):
  - Local Institution - 0038, Maastricht, Limburg
  - Local Institution - 0039, Breda, North Brabant
  - Local Institution - 0277, Leiden, South Holland
  - Local Institution - 0037, Rotterdam, South Holland
- Poland (4):
  - Centrum Medyczne Pratia Poznań, Poznan, Greater Poland Voivodeship
  - Local Institution - 0280, Warsaw, Masovian Voivodeship
  - Local Institution - 0251, Gdask, Pomeranian Voivodeship
  - Local Institution - 0363, Gdansk
- Romania (8):
  - Institutul Regional de Gastroenterologie și Hepatologie Prof. Dr. Octavian Fodor, Cluj-Napoca, Cluj
  - Local Institution - 0111, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Fundeni Clinical Institute, Bucharest
  - Local Institution - 0109, Bucharest
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Institutul Regional de Oncologie, Iași
  - Local Institution - 0108, Ploieşti
- Singapore (4):
  - Local Institution - 0254, Singapore, Central Singapore
  - Local Institution - 0255, Singapore
  - Local Institution - 0252, Singapore
  - Local Institution - 0253, Singapore
- Slovakia (4):
  - Local Institution - 0273, Košice, Košice Region
  - Local Institution - 0274, Trenčín, Trenčín Region
  - Local Institution - 0272, Banská Bystrica
  - Local Institution - 0275, Bratislava
- South Africa (4):
  - Local Institution - 0246, Johannesburg, Gauteng
  - Local Institution - 0241, Pretoria, Gauteng
  - Local Institution - 0240, Soweto, Gauteng
  - Local Institution - 0335, Cape Town, Western Cape
- South Korea (3):
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (7):
  - Local Institution - 0003, Barcelona, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (4):
  - Skånes Universitetssjukhus Lund, Lund, Skåne Län [se-12]
  - Karolinska Universitetssjukhuset Huddinge, Stockholm, Stockholms Län [se-01]
  - Akademiska sjukhuset, Uppsala, Uppsala Län [se-03]
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götalands Län [se-14]
- Switzerland (4):
  - Inselspital Bern, Bern, Canton of Bern
  - Cantonal Hospital St.Gallen, Sankt Gallen, Canton of St. Gallen
  - Ospedale Regionale Bellinzona e Valli, Bellinzona, Canton Ticino
  - Université de Genève, Geneva
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- Turkey (Türkiye) (5):
  - Local Institution - 0284, Stanbul, Istanbul
  - Local Institution - 0283, Adana
  - Local Institution - 0286, Ankara
  - Local Institution - 0287, Ankara
  - Local Institution - 0285, Istanbul
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, England
  - Local Institution - 0014, London, England
  - Royal Marsden Hospital (Chelsea), London, Kensington and Chelsea
  - Guy's & St Thomas' NHS Foundation Trust, London, London, City of
  - Sarah Cannon Research Institute UK, London, London, City of
  - Local Institution - 0235, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07076121.html